CLINICAL TRIAL: NCT03551483
Title: ArtontheBrain: An Inclusive Evidence-based Cognitive Health App for Older Adults to Promote Aging at Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baycrest (Other)
Collaborators: University of Calgary (Other); Sheridan College (Unknown)
Responsible Party: Principal Investigator, Kelly Murphy, Ph.D., C.Psych, Psychologist, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #17-49
Record Dates: First submitted 2018-05-25; First posted 2018-06-11 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-01

CONDITIONS: Cognitive Impairment; Mild Cognitive Impairment; Dementia; Age-related Cognitive Decline; Aging
Keywords: Arts-based Intervention; Mobile Health; Online Recreation
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ArtontheBrain (Experimental): ArtontheBrain application for about 30 to 45 minutes twice per week, over 6 weeks.
  Interventions: Device: ArtontheBrain
- Seniors Online Victoria (Active Comparator): Senior Online Victoria games for about 30 to 45 minutes twice per week, over 6 weeks (https://www.seniorsonline.vic.gov.au/services-information/games), after which they will participate in the ArtontheBrain intervention.
  Interventions: Device: ArtontheBrain; Device: Seniors Online Victoria
- Waitlist Control (Other): The waitlist control group will no treatment for 6 weeks, after which they will six weeks of the ArtontheBrain intervention.
  Interventions: Device: ArtontheBrain

INTERVENTIONS:
Device: ArtontheBrain — The ArtontheBrain intervention has three activities focused on a user selected artwork. The activities promote an in-depth analysis of the artwork and are organized into three activity categories; learn, play, and mingle. In 'learn', the options are to read and/or listen to the curatorial description of the artwork. In 'play', the options are to engage in a word search game, to engage in a visual puzzle game, or to engage in a storytelling game whereby a reminiscence or imaged story can be written. In 'mingle' the options involve social communications about the artwork that include seeing what other comments and seeing how the artwork has been rated by others. The mingle option permits the user to engage only with a select circle of users or to engage with a group of public users.
Device: Seniors Online Victoria — The active control group will use a freely available website, which is updated daily with online games for seniors through an organization called Seniors Online Victoria (https://www.seniorsonline.vic.gov.au/services-information/games).
  Arms: Seniors Online Victoria

SUMMARY:
The research proposed here will evaluate whether a web-based recreation intervention, called ArtontheBrain, has positive health benefits to older adult users. ArtontheBrain incorporates three basic activities; learning (history of the artwork), play (telling stories, solving puzzles) and socializing with other users, either in person or online. It can be used alone, with another person, or in a group. It is modeled after participatory arts-based interventions which studies have shown are associated with health benefits in older adults, such as improved sense of well-being, physical health, decreased risk of dementia, and reduced need for health services. Our study will test ArtontheBrain at research sites and health agencies in Canada, the U.S., and the U.K. with older adults with and without cognitive decline. The study will also examine how well that app can support different user play modalities and whether it can effect positive health outcomes similar to face-to-face arts interventions.

DETAILED DESCRIPTION:
Our project seeks to validate the positive health impacts of a mobile health (mhealth) intervention, called ArtontheBrain; a web-based application (app) aimed at promoting cognitive health in older adults, aging at home, through mentally and socially engaging recreation. The app was created in response to research showing: a) older adults with chronic health conditions experience reduced access to enjoyable recreation due to various barriers (e.g., sensory loss, cognitive decline, mobility limitations, geography and low mood); and b) participatory arts-based recreation is associated with health benefits in seniors (e.g., enhanced well-being, improved physical health, decreased risk of dementia, and reduced use of healthcare resources). There are limited evidence-based solutions for consumers and this clinical validation will provide information about the efficacy of ArtontheBrain in achieving positive health outcomes to guide health practitioners and older adult consumers toward proven products.

Based on quality of life (QOL) benefits for older adults, reported from participatory arts interventions, we hypothesize that engagement with ArtontheBrain will produce similar improvements in QOL in our study participants, driven by specific features of this type of intervention e.g., self-directed, flexible level of complexity, driven by the user. Secondary outcomes hypothesized for engagement with the intervention, include benefits to: active living, aspects of cognition (e.g., attention control, reasoning) and health seeking behaviours. These hypotheses are encouraged by findings from our initial pilot testing which showed improvement in self-perceived health-related QOL and reduced doctor visits in our pilot participants and established proof of principle for the ArtontheBrain with respect to positive user feedback on their experience with this recreation app.

ELIGIBILITY:
Inclusion Criteria:

1. 60 years of age and older.
2. Having normal or corrected to normal vision.
3. Self-reported proficiency in English.
4. Compliance with treatment, over the specified period of 6-weeks.
5. Having experienced:

   1. Age-normal cognitive decline defined as having a Montreal Cognitive Assessment (MoCA) score ≥23 with no functional impairment in Instrumental Activities of Daily Living (iADLs), and no subjective memory complaint;
   2. MCI as defined as having a MoCA score ≤26 with no significant functional impairment in iADLs (e.g., no more than one iADL domain compromised), and report of memory decline by self or family member; or health professional.
   3. Early dementia as defined as MoCA score ≤23 with significant functional impairment in more than one iADLs domain.
6. Having access to a computer (e.g., desktop, laptop, tablet) and internet.

Exclusion Criteria:

1. Significant vision loss (low vision accepted).
2. Non-fluent in English.
3. Major psychiatric disorder.
4. Neurological disorder causing aphasia or causing severe dementia.
5. Motor limitations that prevent independent use of computer technology.
6. Current history of substance abuse.
7. No access to a computer (e.g., desktop, laptop, tablet) or internet.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L | Change from baseline quality of life at 6 week
  The EQ-5D-5L comprises five dimensions on subjectively perceived quality of life in areas of: mobility, self-care, usual activities, pain/ discomfort, and anxiety/ depression. Participants report on a five-point scale whether they have no problems (1), slight problems (2), moderate problems (3), severe problems (4), or extreme problems (5). Then, using a visual analog scale from 0 to 100, individuals are asked to assess their momentary health state (100 indicating the best health state and 0 indicating the worst health state they can imagine).
Short Warwick-Edinburg Mental Well-Being Scale (WEMWBS) | Change from baseline mental wellbeing at 6 weeks
  The Short Warwick-Edinburg Mental Well-Being Scale (WEMWBS) is a 7-item scale designed to measure mental well-being over the previous two weeks. Each statement is positively phrased and measured along a 5-point Likert scale ranging from 1(i.e., never) to 5 (i.e., always). Questions include: "I've been feeling optimistic about the future"; "I've been dealing with problems well"; "I've been able to make up my mind about things".
Short-Form Health Survey (SF-36) | Change from baseline SF-36 score at 6 week
  The Short-Form Health Survey (SF-36) is composed of 36-items that measure health across eight domains including physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/ fatigue, emotional well-being, social functioning, pain and general health.
Stanford Health Care Utilization | Change from baseline health care utilization at 6 week
  The Stanford Chronic Disease Questionnaire Medical Care section evaluates individuals of health care utilization occurring in the previous six months. It comprises 4 items of three types of health care utilization: physician visits, emergency room visits, and hospitalization.

SECONDARY OUTCOMES:
Physical Activity Scale in the Elderly | Change from baseline physical activity at 6 weeks
  The Physical Activity Scale for the Elderly (PASE) is a self-report measure of physical activity in older adults. The PASE comprises 10 items of leisure, household, and occupational activities occurring over the previous seven days. Items on the PASE are scored by multiplying the time spent (i.e., hours per week) or participation (i.e., yes or no) with empirically derived weights. Higher scores indicate higher levels of physical activity.
Social Engagement Survey | Change from baseline social engagement at 6 weeks
  The Social Engagement Survey evaluates an individual's level of social engagement by their social network size, social activities and social support. In the first section, social network size is measured by asking participants to list the names of people in their lives who meet the following criteria: 1) someone with whom you feel close and can talk about personal matters; and 2) someone you have contact with at least once per month. The next section comprises 6-items of social activities measured along a 5-point Likert scale ranging from 1 (i.e., once a year or less) to 5 (i.e., every day or nearly every day) and participants are to report whether they have engaged in that activity in the past year. In the last section, participants are to respond along a 7-point Likert scale ranging from 1 (i.e., very strongly disagree) to 7 (i.e., very strongly agree) on 4-items pertaining to social support.
Alternative Uses Task | Change from baseline score at 6 weeks
  The Alternative Uses Task was designed to evaluate divergent thinking abilities by asking participants to generate as many uses as possible for a given item within the span of one minute. The following six items will be selected from: eyeglasses, shoes, keys, button, wooden pencil and automobile tire. Participant's responses will be recorded and scored for standard measures of divergent thinking including: fluency, flexibility, appropriateness, elaboration and originality
Digit Span Test | Change from baseline score at 6 weeks
  The Forward and Backward Digit Span subtests will be used in the present study as they are associated with central executive functioning in older adults, and with arts-related competence and training. In the forward span subtest, the experimenter will read out a sequence of numbers at the rate of 1 digit/s and the participant will be instructed to recall the numbers in the same order. In the backward span sub test, the participant will recall the numbers in reverse order.
Means-End Problem Solving | Change from baseline score at 6 weeks
  The Means-End Problem Solving (MEPS) test is a standardized measure comprising 10 vignettes, each with a social problem. The participants are given the beginning of the problem and the end of the problem and are asked to describe in detail the middle part of the story out loud. Participants are given as much time as they may need to fully describe their solutions and a general probe is given after each solution described (e.g., Can you think of anything else that you would like to add to this story?) to ensure all details are described and recorded.
Art Engagement Survey | Change in baseline score at 6 weeks
  Engagement in arts-related activities occurring in the previous year will be assessed using the Arts Engagement Survey. Briefly, the survey quantifies art engagement by asking participants questions about participation, learning, work/ volunteering and arts-related membership. For each item, participants are asked whether or not they engaged in that event, and if so, approximately how many days or how many hours they spent engaging in that activity or event.
Life Space Questionnaire (LSQ) | Change in baseline score at 6 weeks
  The Life Space Questionnaire (LSQ) is a brief survey that asks participants to reflect on the extent of their range of travel within and outside the home occurring in the previous three days. It comprises nine items with each item addressing a specific life-space zone. The LSQ is a valid and reliable measure that is useful for establishing the spatial extent for mobility among older adults.
Autobiographical Interview | Change in baseline score at 6 weeks
  The Autobiographical Interview was designed to assess autobiographical memory using a text- based analysis of transcribed protocols. Participants are asked to provide a detailed description of a significant personal event, for example, from early childhood, teenage years, early adulthood, and the past year. Each memory is assessed across free recall, general probe, and specific probe conditions

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Murphy, Ph.D, Principal Investigator — Baycrest Health Sciences
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Background] Noice T, Noice H, Kramer AF. Participatory arts for older adults: a review of benefits and challenges. Gerontologist. 2014 Oct;54(5):741-53. doi: 10.1093/geront/gnt138. Epub 2013 Dec 11. PMID 24336875
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Lyons RA, Perry HM, Littlepage BN. Evidence for the validity of the Short-form 36 Questionnaire (SF-36) in an elderly population. Age Ageing. 1994 May;23(3):182-4. doi: 10.1093/ageing/23.3.182. PMID 8085500
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Davies C, Knuiman M, Rosenberg M. The art of being mentally healthy: a study to quantify the relationship between recreational arts engagement and mental well-being in the general population. BMC Public Health. 2016 Jan 5;16:15. doi: 10.1186/s12889-015-2672-7. PMID 26733272
- [Background] Washburn RA, McAuley E, Katula J, Mihalko SL, Boileau RA. The physical activity scale for the elderly (PASE): evidence for validity. J Clin Epidemiol. 1999 Jul;52(7):643-51. doi: 10.1016/s0895-4356(99)00049-9. PMID 10391658
- [Background] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Levine B, Svoboda E, Hay JF, Winocur G, Moscovitch M. Aging and autobiographical memory: dissociating episodic from semantic retrieval. Psychol Aging. 2002 Dec;17(4):677-89. PMID 12507363
- [Background] Kessels RP, van Zandvoort MJ, Postma A, Kappelle LJ, de Haan EH. The Corsi Block-Tapping Task: standardization and normative data. Appl Neuropsychol. 2000;7(4):252-8. doi: 10.1207/S15324826AN0704_8. PMID 11296689
- [Background] Hester RL, Kinsella GJ, Ong B. Effect of age on forward and backward span tasks. J Int Neuropsychol Soc. 2004 Jul;10(4):475-81. doi: 10.1017/S1355617704104037. PMID 15327726
- [Background] MEDNICK SA. The associative basis of the creative process. Psychol Rev. 1962 May;69:220-32. doi: 10.1037/h0048850. No abstract available. PMID 14472013
- [Background] Murphy KJ, Troyer AK, Levine B, Moscovitch M. Episodic, but not semantic, autobiographical memory is reduced in amnestic mild cognitive impairment. Neuropsychologia. 2008 Nov;46(13):3116-23. doi: 10.1016/j.neuropsychologia.2008.07.004. Epub 2008 Jul 12. PMID 18675285
- [Background] Ritter PL, Stewart AL, Kaymaz H, Sobel DS, Block DA, Lorig KR. Self-reports of health care utilization compared to provider records. J Clin Epidemiol. 2001 Feb;54(2):136-41. doi: 10.1016/s0895-4356(00)00261-4. PMID 11166528
- [Background] Beauchet O, Launay CP, Merjagnan C, Kabeshova A, Annweiler C. Quantified self and comprehensive geriatric assessment: older adults are able to evaluate their own health and functional status. PLoS One. 2014 Jun 26;9(6):e100636. doi: 10.1371/journal.pone.0100636. eCollection 2014. PMID 24968016
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Boot WR, Charness N, Czaja SJ, Sharit J, Rogers WA, Fisk AD, Mitzner T, Lee CC, Nair S. Computer proficiency questionnaire: assessing low and high computer proficient seniors. Gerontologist. 2015 Jun;55(3):404-11. doi: 10.1093/geront/gnt117. Epub 2013 Oct 9. PMID 24107443
- [Background] Fraser KD, O'Rourke HM, Wiens H, Lai J, Howell C, Brett-MacLean P. A Scoping Review of Research on the Arts, Aging, and Quality of Life. Gerontologist. 2015 Aug;55(4):719-29. doi: 10.1093/geront/gnv027. PMID 26179707